CLINICAL TRIAL: NCT03388502
Title: Effectiveness of a Novel Text-Messaging Bot in Patients Undergoing Total Joint Arthroplasty: A Prospective Randomized Controlled Trial
Brief Title: Novel Text-Messaging Bot in Patients Undergoing Joint Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16050101-IRB02
Record Dates: First submitted 2017-12-24; First posted 2018-01-03 (Actual); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-02

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: Total knee arthroplasty; Total hip arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — Spermine Synthase; Educational Status; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text Messaging (SMS) Bot (Experimental): Patients undergoing total joint (hip & knee) arthroplasty will be enrolled in their physician's automated 'Text Messaging (SMS) Bot' in addition to receiving the routine perioperative education and instructions.
  Interventions: Other: Automated Text Messaging (SMS) Bot (intervention group)
- Routine Perioperative Instructions (Active Comparator): Patients undergoing total joint (hip & knee) arthroplasty will receive only their 'Routine Perioperative Instructions'.
  Interventions: Other: Routine perioperative education & teaching (control group)

INTERVENTIONS:
Other: Automated Text Messaging (SMS) Bot (intervention group) — Patients will be enrolled in an 'Automated Text Messaging (SMS) Bot (intervention group)' which is a computer program that sends patients timely reminders, instructions, and videos to help them prepare and recover from surgery.
  Arms: Text Messaging (SMS) Bot
Other: Routine perioperative education & teaching (control group) — Patients will receive the 'Routine perioperative education & teaching (control group)' and will not be enrolled in the physician-specific SMS bot.
  Arms: Routine Perioperative Instructions

SUMMARY:
This study evaluates the addition of an automated physician-specific text-messaging (SMS) bot in patients undergoing total joint arthroplasty. Half of the patients received the traditional perioperative education and instructions (control group), while the other half were enrolled in their physician's SMS bot (intervention group).

DETAILED DESCRIPTION:
In an era of value-based reimbursement and high-volume surgery, the patient experience is becoming increasingly important. Despite publicized efforts to place a greater emphasis on patient-centered care, patients often report poor access to their physician, lack of effective perioperative education, and frustration as their care is commoditized.

A text-messaging (SMS) bot has the potential to help fill some of these voids. Bots are computer programs that are inherently automated to simulate human-like tasks. While a physician may wish he or she could contact each of their patients daily, it would be an impossible undertaking for most. An SMS bot could make daily contact possible by automating it, potentially improving patient education and engagement before and after surgery. Standard SMS has been previously reported to be an effective means for delivering timely information, increasing patient compliance and outcomes (medication adherence, decrease surgical infections with antiseptic showers), and reaching a socioeconomically diverse patient population. Further benefits may be seen with an SMS bot due to its automated capabilities.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria consisted of patients over 18 years of age, scheduled for primary total hip & knee arthroplasty, with smart phone capability, and proficiency in English.

Exclusion Criteria:

* Patients less than 18 years of age, no smart phone capability, poor English proficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J Campbell, MD, Study Director — Rush University Medical Center

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Text Messaging (SMS) Bot | Routine Perioperative Instructions
Started | 76 | 83
Completed | 76 | 83
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: nothing different from the assignment in Participant Flow
Groups:
- Total: Total of all reporting groups
Arm/Group | Text Messaging (SMS) Bot | Routine Perioperative Instructions | Total
Number analyzed (Participants) | 76 | 83 | 159
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 56 | 55 | 111
  >=65 years | 20 | 28 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (8.0) | 60.9 (8.2) | 60.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 71
  Male | 41 | 47 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data not collected.

OUTCOME MEASURES:

1. Primary Outcome: Time Participating in Home-Based Exercises
Description: Stretching, strengthening, and other rehab-specific exercises counted toward their home-based exercises, while walking was excluded.
Time Frame: over a six-week time period after arthroplasty surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Text Messaging (SMS) Bot | Routine Perioperative Instructions
Number analyzed (Participants) | 76 | 83
minutes | 46.4 (17.4) | 37.7 (16.3)

2. Secondary Outcome: Knee Range of Motion
Description: Degrees of flexion and extension of the operative knee will be measured at 6 weeks after surgery.
Time Frame: over a six-week time period after arthroplasty surgery
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Text Messaging (SMS) Bot | Routine Perioperative Instructions
Number analyzed (Participants) | 76 | 83
degrees | 111.9 (13.3) | 108.0 (12.8)

3. Secondary Outcome: Use of Narcotics/Opiates
Description: Medications designated as "narcotics" included any medications that contained: hydrocodone, oxycodone, codeine, morphine, or tramadol. Patients were instructed to record their responses during the same two-hour window each day in a daily diary.
Time Frame: over a six-week time period after arthroplasty surgery
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Text Messaging (SMS) Bot | Routine Perioperative Instructions
Number analyzed (Participants) | 76 | 83
days | 22.5 (13.4) | 32.4 (11.8)

4. Secondary Outcome: Visual Analog Scale (VAS) Mood Score
Description: VAS mood scores were collected from patients on the standard ten-point validated scale. If a patient circled two adjacent numbers on their daily diary, an average of the two numbers were assigned for that day. Minimum score 0. Maximum score 10. Higher score is worse outcome (more pain).
Time Frame: 6 weeks post-operative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text Messaging (SMS) Bot | Routine Perioperative Instructions
Number analyzed (Participants) | 76 | 83
score on a scale | 7.5 (1.8) | 6.5 (1.7)

5. Secondary Outcome: Calls to the Office
Description: The number of patient calls to their physicians office were tracked and recorded.
Time Frame: over a six-week time period after arthroplasty surgery
Measure: Mean (Standard Deviation); unit: number of calls
Arm/Group | Text Messaging (SMS) Bot | Routine Perioperative Instructions
Number analyzed (Participants) | 76 | 83
number of calls | 0.6 (0.8) | 2.6 (3.4)

6. Secondary Outcome: Number of Participants Reporting Satisfaction With Instruction Clarity
Description: Patients were asked to fill out a satisfaction survey six weeks after surgery
Time Frame: over a six-week time period after arthroplasty surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Text Messaging (SMS) Bot | Routine Perioperative Instructions
Number analyzed (Participants) | 73 | 80
Participants | 69 | 38

7. Secondary Outcome: Visits to the Emergency Department (ED)
Description: The number of visits to the ED were tracked and recorded.
Time Frame: over a six-week time period after arthroplasty surgery
Measure: Number; unit: visits
Arm/Group | Text Messaging (SMS) Bot | Routine Perioperative Instructions
Number analyzed (Participants) | 76 | 83
visits | 0 | 4

ADVERSE EVENTS:
Time Frame: 6 weeks.
Description: Does not differ.
Arm/Group | Text Messaging (SMS) Bot | Routine Perioperative Instructions
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/76 | 4/83
Other Adverse Events (participants affected / at risk) | 0/76 | 0/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Text Messaging (SMS) Bot (N=76) | Routine Perioperative Instructions (N=83)
Presentation to the Emergency Department (Musculoskeletal and connective tissue disorders) | 0 (0) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-01-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT03388502/Prot_SAP_000.pdf
  • Informed Consent Form (2017-01-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT03388502/ICF_001.pdf